CLINICAL TRIAL: NCT01014741
Title: Modified Stepwise Ablation Guided by Low Dose Ibutilide in Chronic Atrial Fibrillation
Brief Title: Modified Ablation Guided by Ibutilide Use in Chronic Atrial Fibrillation
Acronym: MAGIC-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor Of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 09-0906
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Catheter Ablation; Complex Fractionate Electrograms
MeSH Terms: conditions — Atrial Fibrillation | interventions — ibutilide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibutilide arm (Experimental)
  Interventions: Drug: Ibutilide
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibutilide — 0.25mg IV ibutilide after PV isolation prior to CFE ablation
  Arms: Ibutilide arm
Drug: Placebo — Placebo after PV isolation prior to CFE ablation.
  Arms: Placebo arm

SUMMARY:
Procedures for ablation of persistent or long lasting atrial fibrillation are frequently long and require extensive ablation. Some electrophysiologists administer the drug ibutilide during these procedures to help organize the fibrillatory activity of the left atrium with the hope that this may shorten the length of the procedure and duration of ablation needed. Currently there is no standardized approach of administering the drug ibutilide during these procedures, thus the investigators cannot be certain that administering this drug does in fact facilitate the procedure. The aim of the MAGIC-AF Trial is to see if administering a standard dose of the drug ibutilide at a standard time in the procedure can allow for a reduction in the ablation procedure time. The investigators hypothesize that administering ibutilide during these procedures will result in a reduction in the procedure and ablation time required.

DETAILED DESCRIPTION:
Definition: Patients with persistent atrial fibrillation will be enrolled in this trial. All patients will be required to be in atrial fibrillation on the day of the procedure. Standard pulmonary vein (PV) isolation will be performed. Patients will be enrolled in the trial if they remain in atrial fibrillation after bi-directional block is obtained in the left and right sided PVs. At this point, patients will be randomized to receive 0.25mg of IV ibutilide or a placebo (normal saline). Patients will then undergo additional ablation with areas of complex fractionate electrograms (CFE) being targeted. The duration of additional CFE ablation and use of additional non-PV ablation (i.e. placement of linear lesions) will be left to the discretion of the operator. Patients will be followed for 1 year. The primary outcome assessed will be freedom from AF at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Males and females will be enrolled in the study.
* Age >18
* Referred for a first ever ablation procedure for symptomatic persistent/permanent AF (only prior ablation of right-sided typical flutter is permitted)
* All patients must understand the requirements of the study and be willing to comply with the post study follow-up requirements.
* Patients must be in atrial fibrillation on the day of the procedure

Exclusion Criteria:

* Any reversible cause of AF (post-surgery, thyroid disorder, etc.)
* Patients with a myocardial infarction or unstable angina in the previous 2 months.
* Patients with a history of rheumatic heart disease
* Patients with congenital heart disease
* Patients with a history of hypertrophic cardiomyopathy
* Patients with LV ejection fraction < 35%
* Class IV congestive heart failure
* Patients who have experienced any cerebral ischemic event, including any TIA in the preceding 1 month.
* Women who are known to be pregnant or have had a positive β-HCG test 7 days prior to procedure.
* Patients with any other significant uncontrolled or unstable medical condition (including uncontrolled clinically significant coagulation disorders).
* Patients whose life expectancy is less than one year.
* History of malignant ventricular arrhythmias or long QT interval (>500msec)
* Prior left-sided cardiac ablation procedure (catheter based or surgical)
* Mental impairment precluding the patient from providing informed consent or completing the appropriate follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Y Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (5):
  - Regional Cardiology Associates, Sacramento, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Of Virginia Health System, Charlottesville, Virginia
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Republic of Korea University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh SM, d'Avila A, Kim YH, Aryana A, Mangrum JM, Michaud GF, Dukkipati SR, Barrett CD, Heist EK, Parides MK, Thorpe KE, Reddy VY. The modified stepwise ablation guided by low-dose ibutilide in chronic atrial fibrillation trial (The MAGIC-AF Study). Eur Heart J. 2016 May 21;37(20):1614-21. doi: 10.1093/eurheartj/ehw003. Epub 2016 Feb 4. PMID 26850076
- [Result] Singh SM, D'Avila A, Kim YH, Aryana A, Mangrum JM, Michaud GF, Dukkipati SR, Callans DJ, Barrett CD, Beras-Jovine MR, Reddy VY. The Modified Ablation Guided by Ibutilide Use in Chronic Atrial Fibrillation (MAGIC-AF) Study: clinical background and study design. J Cardiovasc Electrophysiol. 2012 Apr;23(4):352-8. doi: 10.1111/j.1540-8167.2011.02198.x. Epub 2011 Oct 28. PMID 22034996
- [Derived] Singh SM, d'Avila A, Kim YH, Aryana A, Mangrum JM, Michaud GF, Dukkipati SR, Barrett CD, Heist EK, Parides MK, Thorpe KE, Reddy VY. Termination of persistent atrial fibrillation during pulmonary vein isolation: insight from the MAGIC-AF trial. Europace. 2017 Oct 1;19(10):1657-1663. doi: 10.1093/europace/euw266. PMID 27702847

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibutilide Arm: Ibutilide: 0.25mg IV ibutilide after pulmonary vein isolation (PVI) isolation prior to complex fractionated atrial electrograms (CFAE) ablation
- Placebo Arm: Placebo: Placebo after PVI isolation prior to CFAE ablation.
Period: Overall Study
Arm/Group | Ibutilide Arm | Placebo Arm
Started | 105 | 95
Completed | 94 | 90
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Ibutilide Arm: Ibutilide: 0.25mg IV ibutilide after PVI isolation prior to CFAE ablation.
- Total: Total of all reporting groups
Arm/Group | Ibutilide Arm | Placebo Arm | Total
Number analyzed (Participants) | 105 | 95 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 60 (9) | 60 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 84 | 72 | 156
Ejection Fraction [Mean (Standard Deviation); unit: percent] | 54 (8) | 55 (8) | 54.5 (8)
Left atrial diameter [Mean (Standard Deviation); unit: mm] | 47 (7) | 46 (8) | 46.5 (7.5)
Hypertension [Number; unit: participants]
  yes | 58 | 58 | 116
  no | 47 | 37 | 84
Diabetes [Number; unit: participants]
  yes | 15 | 17 | 32
  no | 90 | 78 | 168
Coronary artery disease [Number; unit: participants]
  yes | 20 | 10 | 30
  no | 85 | 85 | 170
Stroke or transient ischaemic attack [Number; unit: participants]
  yes | 5 | 6 | 11
  no | 100 | 89 | 189
Congestive heart failure [Number; unit: participants]
  yes | 16 | 7 | 23
  no | 89 | 88 | 177
CHA2DS2VASc score [Mean (Standard Deviation); unit: units on a scale] — CHA2DS2VASc Score calculates stroke risk for patients with atrial fibrillation. As CHA2DS2-VASc score increased, rate of thromboembolic event (TE) within 1 year in non-anticoagulated patients with non-valvular AF increased as well. Score of 0 to be low risk for TE events (none seen in cohort at one year), score of 1 intermediate risk (0.6% rate at 1 year), and greater than 1 high risk (3% rate at 1 year).
  units on a scale | 1.6 (1.3) | 1.4 (1.3) | 1.5 (1.3)
Duration of current AF episode [Mean (Standard Deviation); unit: months] | 9 (21) | 10 (22) | 9.5 (21.5)
Duration of longest AF episode [Median (Standard Deviation); unit: month] | 11 (22) | 12 (23) | 11.5 (22.5)
Long-lasting AF [Number; unit: participants]
  yes | 16 | 22 | 38
  no | 89 | 73 | 162
Prior hospitalization for AF [Number; unit: participants]
  yes | 34 | 32 | 66
  no | 71 | 63 | 134
Prior cardioversion [Number; unit: participants]
  yes | 84 | 71 | 155
  no | 21 | 24 | 45
Statin use [Number; unit: participants]
  yes | 35 | 37 | 72
  no | 70 | 58 | 128
ACE inhibitor/ARB use [Number; unit: participants] — ACE, angiotensin-converting enzyme; ARB, angiotensin receptor blocker.
  participants
    yes | 41 | 39 | 80
    no | 64 | 56 | 120
Current B-blocker use [Number; unit: participants]
  yes | 60 | 50 | 110
  no | 45 | 45 | 90
Current anti-arrhythmic drug use [Number; unit: participants]
  yes | 39 | 35 | 74
  no | 66 | 60 | 126
Prior anti-arrhythmic drug use [Number; unit: participants]
  yes | 37 | 36 | 73
  no | 68 | 59 | 127
Current amiodarone use [Number; unit: participants]
  yes | 6 | 10 | 16
  no | 99 | 85 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 Year Freedom From AF / AT
Description: Freedom from atrial arrhythmia after repeat procedures with or without drugs
Time Frame: one year
Population: Ninety-two patients in the ibutilide group and 93 patients in the placebo group remained in AF after study drug administration and underwent CFAE ablation.
Measure: Number; unit: participants
Arm/Group | Ibutilide Arm | Placebo Arm
Number analyzed (Participants) | 92 | 93
participants
  yes | 65 | 62
  no | 27 | 31

2. Secondary Outcome: Procedure Time
Description: Overall procedure duration
Time Frame: at time of the procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ibutilide Arm | Placebo Arm
Number analyzed (Participants) | 105 | 95
minutes | 316 (79) | 321 (81)

3. Secondary Outcome: AF Termination
Description: AF termination with complex fractionated atrial electrograms (CFAE) ablation
Time Frame: at time of the procedure
Measure: Number; unit: participants
Arm/Group | Ibutilide Arm | Placebo Arm
Number analyzed (Participants) | 105 | 95
participants
  yes | 66 | 52
  no | 39 | 43

4. Secondary Outcome: Radiofrequency Ablation Time
Time Frame: at time of the procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ibutilide Arm | Placebo Arm
Number analyzed (Participants) | 105 | 95
minutes | 99 (37) | 104 (42)

ADVERSE EVENTS:
Arm/Group | Ibutilide Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/90
Other Adverse Events (participants affected / at risk) | 0/94 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No